CLINICAL TRIAL: NCT02619929
Title: Assessment of Initial Oral Vinorelbine Dosing Schedules Used for the Treatment of Advanced Non-small-cell Lung Cancer and Metastatic Breast Cancer in Clinical Routine in Germany and Austria (StepUp)
Brief Title: Initial Oral Vinorelbine Dosing Schedules in Clinical Routine in Germany and Austria
Acronym: StepUp
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: DE2015026
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Non-Small-Cell Lung Cancer; Breast Cancer
Keywords: Oral Vinorelbine; Advanced Non-Small-Cell Lung Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vinorelbine oral

SUMMARY:
The aim of this non-interventional study is to assess oral vinorelbine dose schedules (initial dose, dose increase/maintenance/reduction) applied during the initial 8 weeks of treatment under routine conditions in Germany together with the underlying reasons for the respective chosen schedules.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient with regard to the pseudonymized documentation and processing of his/her disease data
* Legally capable male or female NSCLC patient or legally capable female MBC patient; in both situations: ≥ 18 years of age (no upper limit)
* Presence of any of the following two tumor entities:

  * Advanced NSCLC (stage III or IV)
  * Anthracycline- and taxane-resistant MBC (stage IV) in women
* Planned systemic chemotherapy and planned regimen with oral vinorelbine in any palliative setting (decision on treatment must have been made before inclusion in this study); included treatments:

  * Monotherapy or any combination therapy with oral vinorelbine
  * Inclusion of patients with hybrid-treatment involving i.v. and oral vinorelbine in one treatment cycle is allowed

Exclusion Criteria:

* Presence of any contraindication with regard to oral vinorelbine treatment (and with regard to i.v. vinorelbine in case of hybrid-treatment) according to the respective Summary of Product Characteristics (SmPC)
* Oral vinorelbine based palliative treatment already ongoing or planned oral vinorelbine starting dose of >60 mg/m2
* Presence of a Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 2
* Simultaneous participation in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Palliative patients with advanced non-small-cell lung cancer (NSCLC, stage III and IV) or anthracycline/taxane-resistant metastatic breast cancer (MBC, stage IV)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Rate of patients with oral vinorelbine dose increase from ≤60 to ≥80 mg/m² during the course of the study | 8 weeks of treatment
  The outcome will be calculated together with its negative (i.e. the rate of patients without such dose increase). Reasons for increasing and for not increasing the dose will be analyzed.

SECONDARY OUTCOMES:
Body weight | Baseline and 8 weeks of treatment
  Body weight [kg] at baseline and changes during the study
Body mass index | Baseline and 8 weeks of treatment
  Body mass index [kg/m^2] at baseline and changes during the study
Body surface area | Baseline and 8 weeks of treatment
  Body surface area [m^2] at baseline and changes during the study
ECOG performance status | Baseline and 8 weeks of treatment
  ECOG performance status [grades 0-5] at baseline and changes during the study
Treatment regimen | Baseline
  Frequency analysis of planned treatment regimens (monotherapy, combination, combination compounds) at baseline. Reasons for choosing the treatment regimen will be analyzed.
Treatment changes | 8 weeks of treatment
  Frequency analysis of dose changes and of the underlying reasons
Relationships between oral vinorelbine dose increases and patient and disease characteristics | Baseline and 8 weeks of treatment
  Generalized linear mixed model with the variable "dose increase" as binary response variable
Assessment of initial tumor response (based on clinical or imaging assessment) | 8 weeks of treatment
Patient's quality of life | Baseline and 8 weeks of treatment
  Evaluation of the patient's quality of life [Short Form (SF)-12]
Patient's treatment satisfaction | 8 weeks of treatment
  Evaluation of the patient's treatment satisfaction [Cancer Therapy Satisfaction Questionnaire (CTSQ)]
Physician's treatment satisfaction | 8 weeks of treatment
  Evaluation of the physician's treatment satisfaction [5 point scale]
Adverse drug reactions | 8 weeks of treatment
  Evaluation of adverse drug reactions using CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (56):
- Austria (7):
  - Braunau am Inn
  - Graz
  - Innsbruck
  - Klagenfurt
  - Vienna
  - Villach
  - Vöcklabruck
- Germany (49):
  - Aachen
  - Altötting
  - Amberg
  - Bad Nauheim
  - Ballenstedt
  - Berlin
  - Bielefeld
  - Chemnitz
  - Cologne
  - Dessau
  - Donauwörth
  - Eggenfelden
  - Erbach im Odenwald
  - Erfurt
  - Frankfurt am Main
  - Göppingen
  - Greifswald
  - Güstrow
  - Halle
  - Hanover
  - Heppenheim an der Bergstrasse
  - Homburg
  - Karlsruhe
  - Kiel
  - Kulmbach
  - Lich
  - Lostau
  - Ludwigsburg
  - Lübeck
  - Mainz
  - Mannheim
  - Marktredwitz
  - Memmingen
  - Munich
  - Münster
  - Offenbach
  - Offenburg
  - Ostfildern
  - Regensburg
  - Saarbrücken
  - Schwandorf in Bayern
  - Solingen
  - Stolberg
  - Villingen-Schwenningen
  - Waltershausen
  - Weinheim
  - Werdau
  - Wesel
  - Winnenden